CLINICAL TRIAL: NCT00879983
Title: An Open Label, Randomized, Crossover Study To Estimate The Pharmacokinetics And Evaluate The Safety Following A Single Dose Of Azithromycin 2g Extended-Release Powder For Oral Suspension With A 3-Day Dosing Regimen Of Azithromycin 500mg Tablet In Chinese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A0661179
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Volunteers
Keywords: azithromycin, pharmacokinetics
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Will accept azithromycin ER first, after at least 14 days washout, then accept azithromycin tablet.
  Interventions: Drug: azithromycin (Zithromax)
- Group 2 (Other): Will accept azithromycin tablet first, after at least 14 days washout, then accept azithromycin ER .
  Interventions: Drug: azithromycin (Zithromax)

INTERVENTIONS:
Drug: azithromycin (Zithromax) — 1. a single dose of azithromycin ER 2g
  2. 3-day regimen of azithromycin tablet 500mg
  Other Names: Zithromax
  Arms: Group 1
Drug: azithromycin (Zithromax) — 1. 3-day regimen of azithromycin tablet 500mg
  2. a single dose of azithromycin ER 2g
  Other Names: Zithromax
  Arms: Group 2

SUMMARY:
The purpose of this study is to estimate the pharmacokinetics and evaluate the safety following a single dose of azithromycin 2g extended-release powder for oral suspension with a 3-day dosing regimen of azithromycin 500mg tablet in Chinese healthy male subjects. This study data will be used to support azithromycin NDA in China.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* Male.
* 18-45 years old.
* BMI 17.5-30.5 kg/m2.

Exclusion Criteria:

* Alcohol, drug, smoke user.
* Sensitive to macrolide antibiotics class drug, parn or heparin-induced thrombocytopenia.
* Severe medical or psychiatric condition or laboratory abnormality.
* Blood donation.
* 12-ECG abnormal.
* Treatment with study drug; clinically significant.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
AUC inf (if data permit) and AUC last of azithromycin | 2 months

SECONDARY OUTCOMES:
AUC 24, Cmax, Tmax, t1/2 of azithromycin | 2 months
vital signs, 12-lead ECG, laboratory tests and adverse events. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Shanghai, China

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661179&StudyName=An%20Open%20Label%2C%20Randomized%2C%20Crossover%20Study%20To%20Estimate%20The%20Pharmacokinetics%20And%20Evaluate%20The%20Safety%20Following%20A%20Single%20Dose%20Of%20Azith